CLINICAL TRIAL: NCT02664688
Title: Lumbar Stabilization Exercises vs Flexor Exercises in Patients With Chronic Low Back Pain and Degenerative Spondylolisthesis
Brief Title: Lumbar Stabilization Exercises vs Flexor Exercises in Degenerative Spondylolisthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Tania Ines Nava-Bringas, MSc; MD, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19/15
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2018-03

CONDITIONS: Degenerative Spondylolisthesis; Chronic Low Back Pain
Keywords: spondylolisthesis; low back pain; stabilization exercise
MeSH Terms: conditions — Spondylolisthesis; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar stabilization exercises (Experimental): Home exercise program to perform daily for 6 months
  Interventions: Other: Lumbar stabilization exercises
- Flexor Exercises (Active Comparator): Home exercise program to perform daily for 6 months
  Interventions: Other: Flexor exercises

INTERVENTIONS:
Other: Lumbar stabilization exercises — The home-exercise program included an initial phase, with use of therapeutic heat via a hot pack for 15 minutes at the lumbosacral region, stretching exercises of the thoracolumbar fascia, hip flexors, hamstrings plus the stabilization exercises to encourage stabilizing motor patterns and determine the neutral position of the spine, with the target in control of transversus and internal oblique abdominis, multifidus, pelvic floor muscles, and diaphragmatic breathing control. Progression stages included hot packs, stretching exercises, and lateral, anterior bridges, leg raises in supine position, and arm and leg lifts in quadruped position ("bird-dog")
  Arms: Lumbar stabilization exercises
Other: Flexor exercises — The home-exercise program included a hot pack for 15 minutes and flexor exercises routine
  Other Names: Williams exercises
  Arms: Flexor Exercises

SUMMARY:
The purpose of this study is to compare the effectiveness of pain control and functional improvement in patients with degenerative spondylolisthesis treated with "lumbar stabilization exercises" vs "flexor exercises (williams exercises)"

DETAILED DESCRIPTION:
This study is a randomized controlled trial in patients with the diagnosis of degenerative spondylolisthesis.

To date, it is known that lumbar stabilization exercises are an effective treatment option in controlling pain and improving function in patients with degenerative spondylolisthesis based on previous studies, but it is not known if is this a better treatment that another exercises routine for chronic LBP (Low Back Pain).

The purpose is to compare the effectiveness on pain control and functional improvement of "lumbar stabilization exercises" vs "flexor exercises (williams exercises)".

All clinical evaluations are performed by a single physician who is blinded to the exercises, and include a full medical history, physical examination, and x-ray measurement.

After initial evaluation, patients are given a sealed envelope containing the treatment (by simple randomization assigned by the investigator). The envelope is opened by the physical therapist which schedules a monthly session and verify the correct execution of each exercise. Each patient receives a sheet with instructions of the exercises to continue daily at home.

Scales to assess pain and function will be recorded at baseline, 4 weeks, 3 months and at 6 months to complete the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative spondylolisthesis at L4-L5 and chronic LBP with or without radicular pain
* Attending the Spinal Rehabilitation Service of the National Institute for Rehabilitation (Mexico City).
* Without previous treatment
* Agree to participate through informed consent.

Exclusion Criteria:

* History of lumbar surgery,
* Rheumatic diseases: Rheumatoid Arthritis, Lupus Erythematosus Systemic, Fibromyalgia, etc.
* Cauda equine symptoms,
* Ischemic heart disease
* Diabetic polyneuropathy
* Illiterate

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in Pain (VAS) | At baseline, 4 weeks, 3 months and 6 months
  Visual Analog Scale (VAS), considering "no pain" to be at 0mm, and 100mm to be "unbearable pain."
Change in Disability (The Roland Morris Scale) | At baseline, 4 weeks, 3 months and 6 months
  The Roland Morris Scale: a self-administered questionnaire consisting of 24 items. The total score can range from 0 (no disability) to 24 (maximum disability)

SECONDARY OUTCOMES:
Change in use of analgesics | At baseline, 4 weeks, 3 months and 6 months
  Total number of days consuming analgesics in the 30 days prior to the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: TANIA I NAVA-BRINGAS, MSc, Principal Investigator — Instituto Nacional de Rehabilitacion
Locations (1):
- INRMexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nava-Bringas TI, Hernandez-Lopez M, Ramirez-Mora I, Coronado-Zarco R, Israel Macias-Hernandez S, Cruz-Medina E, Arellano-Hernandez A, Leon-Hernandez SR. Effects of a stabilization exercise program in functionality and pain in patients with degenerative spondylolisthesis. J Back Musculoskelet Rehabil. 2014;27(1):41-6. doi: 10.3233/BMR-130417. PMID 23948848
- [Result] Vasquez-Rios JR, Nava-Bringas TI. [Lumbar stabilization exercises]. Cir Cir. 2014 May-Jun;82(3):352-9. Spanish. PMID 25238480
- [Derived] Nava-Bringas TI, Romero-Fierro LO, Trani-Chagoya YP, Macias-Hernandez SI, Garcia-Guerrero E, Hernandez-Lopez M, Roberto CZ. Stabilization Exercises Versus Flexion Exercises in Degenerative Spondylolisthesis: A Randomized Controlled Trial. Phys Ther. 2021 Aug 1;101(8):pzab108. doi: 10.1093/ptj/pzab108. PMID 33792726